CLINICAL TRIAL: NCT01238328
Title: Hematopoietic Stem Cell Transplantation for Mucopolysaccharidosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HORCSCT-0906
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Mucopolysaccharidosis
Keywords: Mucopolysaccharidosis; HSCT
MeSH Terms: conditions — Mucopolysaccharidoses | interventions — Transplantation Conditioning; Cyclophosphamide; Antilymphocyte Serum; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation (Experimental)
  Interventions: Drug: Conditioning regimen; Drug: Graft-versus-host disease (GVHD) prophylaxis; Procedure: Stem Cell Transplantation

INTERVENTIONS:
Drug: Conditioning regimen — For sibling full match:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  For other related full match, sibling or other related with one antigen mismatch and umbilical cord blood:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  * Antithymocyte globulin (ATG) rabbit (Thymoglobulin) 10 mg/kg or ATG horse (Atgam) 40 mg/kg
  For haploidentical:
  * Busulfan 16 mg/kg >5year - 20 mg/kg <5year po
  * Cyclophosphamide 200 mg/kg iv
  * Fludarabine 160 mg/m^2
  Other Names: Endoxan; Antithymocyte globulin (ATG) rabbit : Thymoglobulin; Antithymocyte globulin (ATG) horse : Atgam
Drug: Graft-versus-host disease (GVHD) prophylaxis — * Cyclosporin A 1.5 mg/kg/day iv from -2, then 3 mg/kg/day iv (from +7 in peripheral blood stem cell transplant (PBSCT) and +11 in Bone marrow transplantation or Umbilical Cord Blood (UCB) transplantation) then 9 mg/kg/day po
  * 10 mg/m^2 iv day +1 then 6 mg/m^ iv day +3 and +6 (Not for UCBT)
  Other Names: MTX
Procedure: Stem Cell Transplantation — Patients undergoing Hematopoietic Stem Cell Transplantation from one of below source:
  1. Sibling full match
  2. Other related full match
  3. Sibling or other related with 1 mismatch antigen
  4. Cord Blood
  5. Haploidentical
  Other Names: HSCT

SUMMARY:
The purpose of this study is to evaluate the efficacy and side effects of donor hematopoietic cells using chemotherapy regimen without total-body irradiation in children undergoing a hematopoietic stem cell transplant for Mucopolysaccharidosis. The blood stem cells will be derived from either related donor or unrelated umbilical cord blood or haploidentical donor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mucopolysaccharidosis type 1, 6 and 7 confirm by leukocyte enzyme assay
* Age up to 8 year old
* Have suitable donor

Exclusion Criteria:

* Creatinine clearance ≤ 40ml/min/1.73m^2
* Bilirubin ≥ 3mg/dL
* SGPT ≥ 500 U/L
* Current severe infection
* Evidence of CNS involvement
* Morbidity such as blindness or deafness

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival and Progressive Free Survival in patient with Mucopolysaccharidosis who receive allogeneic Hematopoietic stem cell transplantation (HSCT) | 1 year

SECONDARY OUTCOMES:
One year overall survival after allogeneic hematopoietic stem cell transplantation (HSCT) | 1 year
One year Progressive Free Survival after allogeneic hematopoietic stem cell transplantation (HSCT) | 1 year
Transplantation Related Mortality (TRM) after allogeneic hematopoietic stem cell transplantation (HSCT) | 1 year
Acute and chronic Graft-versus-host disease (GVHD) rate after allogeneic hematopoietic stem cell transplantation (HSCT) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology-Oncology & SCT Research Center, Teharn, Tehran Province, Iran